CLINICAL TRIAL: NCT01727180
Title: Pruritus in Patients With Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 100047-E
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Kidney Failure, Chronic; Pruritus
MeSH Terms: conditions — Kidney Failure, Chronic; Pruritus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic kidney disease
  Interventions: Other: Questionnaire based on the McGill Pain Questionnaire

INTERVENTIONS:
Other: Questionnaire based on the McGill Pain Questionnaire — Interview questionnaire based on the short form of the McGill Pain Questionnaire

SUMMARY:
We believe that knowing characteristics of uremic pruritus is the foundation to investigate its pathophysiology and offer better skin care for patients with chronic kidney disease. We therefore conducted this cross-sectional study to evaluate the characteristics of uraemic pruritus.

ELIGIBILITY:
Inclusion Criteria:

* Adults older than 20 years old, with CKD stage 3 to 5D, with symptoms of pruritus.

Exclusion Criteria:

* Patients who refused to answer the questionnaire or unable to understand the contents of the questionnaire.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CKD stage 3 to 5D, followed-up in the Far Eastern Memorial Hospital
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hon-Yen Wu, MD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chronic Kidney Disease
Started | 108
Completed | 108
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chronic Kidney Disease
Number analyzed (Participants) | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 53

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS)
Description: A visual analog scale (VAS) measuring the general severity of pruritus was reported from 0 to 10 (0 = no pruritus, 10 = worst pruritus imaginable
Time Frame: Once at the entry of the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chronic Kidney Disease
Number analyzed (Participants) | 108
units on a scale | 3.35 (2.27)

ADVERSE EVENTS:
Arm/Group | Chronic Kidney Disease
Serious Adverse Events (participants affected / at risk) | 0/108
Other Adverse Events (participants affected / at risk) | 0/108

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No